CLINICAL TRIAL: NCT03189069
Title: Real-World Comparisons of Bleeding Among Novel Oral Anticoagulant (NOAC)-Naïve Non-Valvular Atrial Fibrillation (NVAF) Patients With Medicare Advantage Coverage, Who Newly Initiated Novel Oral Anticoagulation Therapies or Were Treated With Warfarin
Brief Title: A Real-World Comparison of Safety and Effectiveness of Novel Oral Anti-Coagulant (NOAC) Naïve and Warfarin Naïve Non-Valvular Atrial Fibrillation (NVAF) Patients With Medicare Advantage Coverage
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-583
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients prescribed apixaban
  Interventions: Drug: Apixaban
- Patients prescribed dabigatran
  Interventions: Drug: Dabigatran
- Patients prescribed rivaroxaban
  Interventions: Drug: Rivaroxaban
- Patients prescribed warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Treatment for NVAF patients
  Groups: Patients prescribed apixaban
Drug: Dabigatran — Treatment for NVAF patients
  Groups: Patients prescribed dabigatran
Drug: Rivaroxaban — Treatment for NVAF patients
  Groups: Patients prescribed rivaroxaban
Drug: Warfarin — Treatment for NVAF patients
  Groups: Patients prescribed warfarin

SUMMARY:
The primary purpose of this study is to evaluate the risk of major bleeding and stroke/systemic embolism (SE) among novel oral anti-coagulant (OAC) naïve and warfarin naïve Medicare Advantage patients with non-valvular atrial fibrillation (NVAF) treated with apixaban, dabigatran, rivaroxaban, or warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Had at least 1 pharmacy claim for warfarin, apixaban, dabigatran, or rivaroxaban during the identification period (01-Jan-2013 through 31-Dec-2015)
* Had continuous health plan enrollment with medical and pharmacy benefits for 6 months pre-index date (baseline period)
* Had continuous health plan enrollment with medical and pharmacy benefits for at least 1 month following index date
* Had at least 1 medical claim for atrial fibrillation any time before or on index date

Exclusion Criteria:

* Had medical claims with a diagnosis code for rheumatic mitral valvular heart disease, mitral valve stenosis or heart valve replacement/transplant during the 6-month baseline period
* Had medical claims with a diagnosis code for dialysis, kidney transplant, or end-stage chronic kidney disease during the 6 month baseline period
* Had medical claims indicating a diagnosis of venous thromboembolism during the 6-month baseline period
* Had claims indicating a diagnosis or procedure code of hip or knee replacement surgery within 6 weeks prior to the index date
* Had claims for a diagnosis or procedure code for reversible atrial fibrillation
* Had medical claims indicating pregnancy during the study period
* Had a pharmacy claim for warfarin, apixaban, dabigatran, edoxaban, or rivaroxaban during the 6-month baseline period
* Had > 1 oral anticoagulant prescription claim on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the MORE Registry according to the inclusion/exclusion criteria. Four different cohorts will be evaluated: patients who were prescribed warfarin, apixaban, dabigatran or rivaroxaban. Only users of oral anticoagulant treatment from January 1, 2013 to January 1, 2016 will be included in this study.
Sampling Method: Probability Sample
Enrollment: 36000 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Major bleeding | 36 months

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx